CLINICAL TRIAL: NCT07103447
Title: A Prospective, Multicenter, Single-Arm Study of AK112 in Combination With Albumin-Bound Paclitaxel and Carboplatin as Neoadjuvant Treatment for Triple-Negative Breast Cancer
Brief Title: Prospective Multicenter Single-arm Trial: AK112 + Nab-paclitaxel/Carboplatin Neoadjuvant for TNBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shuangyue Liu (Other)
Responsible Party: Sponsor-Investigator, Shuangyue Liu, Chief physician, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WestChinaL112
Record Dates: First submitted 2025-01-17; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer - Female
Keywords: AK112 combining chemothrapy, neoadjuvant therapy, TNBC
MeSH Terms: interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AK112 combining Nab-paclitaxel and carboplatin (Experimental)
  Interventions: Drug: AK112, Carboplatin, Paxlitaxel

INTERVENTIONS:
Drug: AK112, Carboplatin, Paxlitaxel — The combination of AK112, a platinum-based chemotherapy agent, and Paxlitaxel is administered every three weeks as a neoadjuvant treatment for triple-negative breast cancer. After completing six cycles of this regimen, the participant undergoes surgical treatment.

SUMMARY:
This prospective, multicenter, single-arm clinical study aims to evaluate the efficacy and safety of AK112 in combination with albumin-bound paclitaxel and carboplatin as neoadjuvant treatment in adult women with early or locally advanced triple-negative breast cancer (TNBC). The study seeks to address the pathological complete response (pCR) rate, objective response rate (ORR), breast conservation rate, and invasive disease-free survival (iDFS) following treatment with AK112 combined with albumin-bound paclitaxel and carboplatin in early or locally advanced TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary Participation and Informed Consent: The participant voluntarily agrees to join this clinical trial, signs a written informed consent form, understands the study, and is willing to comply with all trial procedures.
2. Eligibility by Age and Gender: Female participants aged ≥18 years and ≤75 years on the day of signing the informed consent form.
3. Pathological Confirmation of Disease: Histopathologically confirmed diagnosis of T1-4N0-3M0 (except for T1N0M0) triple-negative invasive breast cancer, defined as negative for estrogen receptor (ER) and progesterone receptor (PgR) (immunohistochemistry: ER, PR < 1%), and human epidermal growth factor receptor 2 (HER2) (immunohistochemistry HER2 "0~1+"; or immunohistochemistry HER2 "2+" with no amplification on HER2 FISH gene testing).
4. Measurable Lesion: At least one lesion measurable according to RECIST v1.1 criteria. Participants diagnosed at an external institution agree to provide archived or freshly obtained tumor tissue samples (formalin-fixed paraffin-embedded [FFPE] tissue blocks or at least 25 unstained tumor tissue slides) for pathology review.
5. Planned Surgical Treatment: Participants are scheduled to undergo definitive surgical resection of breast cancer, including either breast-conserving surgery or mastectomy, along with sentinel lymph node (SN) biopsy or axillary lymph node dissection (ALND), and are planned to receive neoadjuvant chemotherapy.

Exclusion Criteria:

1. Prior Anti-Cancer Treatments.
2. Received systemic anti-cancer treatment, including chemotherapy, radiotherapy, immunotherapy, targeted therapy (within 2 weeks for small molecule targeted therapies), or biological agent treatment within 4 weeks before enrollment.
3. Received palliative local treatments within 2 weeks before enrollment.
4. Received systemic non-specific immune modulatory treatments (e.g., interleukins, interferons, thymopeptides) within 2 weeks before enrollment.
5. Received traditional Chinese medicine or Chinese patent medicines with anti-cancer indications within 2 weeks before enrollment.
6. Prior PD-1/PD-L1 Treatment.
7. Previously received treatment with PD-1 inhibitors or PD-L1 inhibitors.
8. Concurrent Participation in Other Clinical Studies.
9. Currently participating in another clinical study, unless it is an observational, non-interventional study or the follow-up period of an interventional study.
10. History of Other Malignancies:

(1) Has a history of other malignant tumors within 5 years prior to enrollment or concurrently, except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, and thyroid cancer.

(2) Active Autoimmune Diseases: Has active autoimmune diseases that required systemic treatment (such as corticosteroids) within 2 years before enrollment, or has autoimmune diseases that the investigator judges may recur or require planned treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR | After surgery, within an average of 2 weeks
  pathological complete response

SECONDARY OUTCOMES:
ORR | Two weeks after completing 6 cycles of neoadjuvant therapy (each cycle is 21 days)
  After complete 6 cycles of neoadjuvant chemotherapy in combination with AK112

IPD SHARING:
Plan to Share IPD: No
The informed consent documents approved by the ethics committee did not cover broad data sharing.